CLINICAL TRIAL: NCT04320225
Title: A Prospective Observational Study: Connection Between Vitamin D Level and the Efficacy of Dexamethasone in Immune Thrombocytopenia
Brief Title: Connection Between Vitamin D Level and the Efficacy of Dexamethasone in Immune Thrombocytopenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor, Shandong University
Other Study IDs: ITP-vitamin D(observational)
Record Dates: First submitted 2020-03-21; First posted 2020-03-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lower vitamin D level group: The vitamin D level is lower than 20 nmol/L.
  Interventions: Drug: Dexamethasone
- Higher vitamin D level group: The vitamin D level is higher than 20 nmol/L.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — HD-DXM (orally at 40 mg daily for 4d )

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. The objective is to find out if there is a connection between vitamin D level and the efficacy of dexamethasone for the treatment of adults with newly-diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a prospective, observational，non-randomized control trial of 60 ITP adult patients. Dexamethasone (given orally at a dose of 40 mg per day for 4 days, two-cycles with an interval of 10 days) will be used in the target patients. Vitamin D level will be detected before the utilization of treatment measures. Depend on the vitamin D level, the patients will be divided into 2 groups(higher vitamin D level group and lower vitamin D level group).Platelet count, bleeding and other symptoms were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

Corresponding to the diagnostic criteria for immune thrombocytopenia Newly diagnosed ITP patients To show a platelet count <30 * 10^9/L, and with bleeding manifestations Willing and able to sign written informed consent

Exclusion Criteria:

Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit; Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit; Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study; Current HIV infection; Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia) Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period; Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test; Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed ITP patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Sustained response to ITP treatments | 3 months after treatment started
  Percentage of patients maintaining PLT count over 30*10^9/L without bleeding